CLINICAL TRIAL: NCT05635786
Title: Early Successful Recanalization After Intravenous Thrombolysis With Tenecteplase Versus Alteplase in Distal Vessel Occlusion Strokes
Brief Title: Early Recanalization After Intravenous Thrombolysis With Tenecteplase Versus Alteplase in Distal Vessel Occlusion Strokes
Acronym: DISTAL-IVT
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Sud Francilien (Other)
Responsible Party: Sponsor
Other Study IDs: 2022/0037
Record Dates: First submitted 2022-11-23; First posted 2022-12-02 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Acute Distal Vessel Occlusion Stroke
Keywords: Acute; occlusion; recanalization; tenecteplase; alteplase; thrombolysis; ischemic; stroke-distal
MeSH Terms: conditions — Bites and Stings; Ischemia | interventions — Tissue Plasminogen Activator; Tenecteplase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Alteplase (ALT): Patients with distal vessel occlusion stroke treated with alteplase (from March 2016 to February 2018)
  Interventions: Drug: Alteplase (0.9mg/kg)
- Tenecteplase (TNK): Patients with distal vessel occlusion stroke treated with tenecteplase (from March 2018 to February 2020)
  Interventions: Drug: Tenecteplase (0.25mg/kg)

INTERVENTIONS:
Drug: Alteplase (0.9mg/kg) — Intravenous thrombolysis with Alteplase (0.9 mg/kg, maximum 90 mg) with 10% of the dose given as a bolus followed by an infusion lasting 60 minutes.
  Groups: Alteplase (ALT)
Drug: Tenecteplase (0.25mg/kg) — Intravenous thrombolysis with Tenecteplase (0.25mg/kg, maximum 25 mg) with 100% of the dose given as a bolus.
  Groups: Tenecteplase (TNK)

SUMMARY:
The purpose of this monocentric retrospective study is to compare, in patients with acute distal vessel occlusion stroke, the early rates of successful recanalization in patients treated with Alteplase (ALT) versus Tenecteplase (TNK), based on a retrospective analysis of magnetic resonance imaging (MRI) performed early after IVT.

DETAILED DESCRIPTION:
Early rates of successful recanalization (SR) of distal vessel occlusions (DVO) following intravenous thrombolysis (IVT) between alteplase (ALT) and tenecteplase (TNK) are poorly known.

From March 2016 to February 2020, consecutive stroke patients hospitalized in the stroke unit of the Sud-Francilien Hospital with DVO identified on baseline MRI and suitable for IVT but not for mechanical thrombectomy will be included. In our stroke unit, patients were treated with ALT, 0.9 mg/kg from March 2016 to February 2018 and then with TNK, 0.25 mg/kg from March 2018 to December 2023. MRI was controlled 1-2 hours within IVT (MRI-2). Early recanalization was assessed on an adapted Arterial Occlusion Lesion (AOL) scale, SR being defined as AOL 2/3 scores on MRI-2. The rate reduction of thrombus length (TL) when thrombus persisted, the IVT response threshold of TL and the infarct size evolution were also assessed. In the present study, the investigators sought to compare early rates of SR between the two lytics, based on a retrospective analysis of magnetic resonance imaging (MRI) performed early after IVT.

ELIGIBILITY:
Inclusion Criteria:

* Age≥ 18 years.
* Acute ischemic stroke (visible on DWI, but not visible on FLAIR) on initial MRI associated with distal arterial occlusion as defined below:

  * A distal occlusion of the M2 segment of the middle cerebral artery (MCA)
  * Occlusion (regardless of location) of a non-dominant M2 branch of the MCA
  * Occlusion of the M3 segment of the MCA.
  * Occlusion of the A2 or A3 segment of the anterior cerebral artery (ACA)
  * Occlusion of the P2 or P3 branch of the posterior cerebral artery (PCA).
  * A proximal M2-MCA or proximal P1-PCA occlusion may also be included if not eligible for mechanical thrombectomy, especially if the initial NIHSS score is low (<5).
  * Distal arterial occlusion is identified by MRI either on the TOF (Time of Flight)-ARM sequence and/or on the presence of a thrombus (Susceptibility Vessel sign, SVS) on the SWAN sequence,
* IVT by ALT or TNK within 4H30 after onset of symptoms,
* Early brain MRI performed 1 to 2 hours after IVT (MRI n°2),
* Good quality MRI (absence of motion artifact interfering with interpretation) with availability of DWI, FLAIR, TOF-MRA and SWAN sequences.

Exclusion Criteria:

- Patients informed of the study who objected to the collection of their data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a monocentric retrospective study (Sud-Francilien Hospital (SFH), Corbeil-Essonnes, France) based on a stroke registry prospectively gathered.
  From March 2016 to February 2020, consecutive patients with acute ischemic stroke (AIS) assessed on brain MRI and treated with IVT alone who fulfilled the following criteria will be included: 18 years or older; evidence of an AIS on acute MRI (MRI-1) associated with a distal vessel occlusion as defined below; IVT within 4h30 of symptoms onset; availability of a post-IVT MRI within 1-2 hours (MRI-2); good quality of MRI sets including SWAN images.
Sampling Method: Probability Sample
Enrollment: 319 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2024-11-21 (Actual); Study Completion 2024-11-21 (Actual)

PRIMARY OUTCOMES:
Early successful recanalization rate | Between 1 and 2 hours after IVT
  Early successful recanalization rate defined by an Arterial Occlusive Lesion (AOL) scale grade 2 or 3 on MRI-2 performed between 1 and 2 hours after IVT.

SECONDARY OUTCOMES:
Early complete recanalization rate | Between 1 and 2 hours after IVT
  Early complete successful recanalization rate defined by an Arterial Occlusive Lesion (AOL) scale grade 3 on MRI-2 performed between 1 and 2 hours after IVT.
Thrombus length change | Between 1 and 2 hours after IVT
  Thrombus length (TL) was approximated by measuring the susceptibility vessel sign (SVS) on the susceptibility weight angiography (SWAN) sequence.
  TL were measured in the 3 spatial planes, the higher value being retained. When thrombus persisted on MRI-2, TL reduction was assessed as follows : (MRI-1 length - MRI-2 length)/MRI-1 length X 100.
Evolution of cerebral infarct volume | Between 1 and 2 hours after IVT
  Volume of the ischemic lesion will be assessed on the diffusion-weighted imaging (DWI) sequence using an automated software (Olea software).
  This evolution of cerebral infarct volume will be calculated as follows : DWI MRI volume n°2 - initial DWI MRI volume.
Rates of early post-thrombolysis intracerebral hemorrhage | Between 1 and 2 hours after IVT
  Rates of early post-thrombolysis intracerebral hemorrhage on MRI-2 (performed at 1 to 2h after IVT) according to the Heidelberg classification (Kummer et al, Stroke 2015)
Very early clinical modification | Between 1 and 2 hours after IVT
  Very early neurological modification was assessed as follows : baseline NIHSS -NIHSS at H1.
  Very early clinical improvement (VENI) was defined as baseline NIHSS -NIHSS at H1. ≥4, or NIHSS H1=0.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Sud Francilien, Corbeil-Essonnes, France, France

IPD SHARING:
Plan to Share IPD: No